CLINICAL TRIAL: NCT01631084
Title: A Multicentre Randomized Program to Compare the Effect of the Joint Asia Diabetes Evaluation (JADE, Structured Care) Versus the DIAbetes MONitoring Database (DIAMOND, Usual Care) Programs in Type 2 Diabetes in the Asia Pacific Region
Brief Title: Comparing the Effect of Structured Care Versus Usual Care in Type 2 Diabetes Patients Across the Asia Pacific Region
Acronym: AP-JD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia Diabetes Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2012.199-T
Record Dates: First submitted 2012-06-27; First posted 2012-06-28 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Diabetes
Keywords: Diabetes; Structured care
MeSH Terms: conditions — Diabetes Mellitus | interventions — Diamond

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JADE (Experimental): Patients randomized to the JADE group will be followed according to protocol-driven diabetes care based on their individual risk levels, using a web-based disease management program. In addition to their annual comprehensive assessments at baseline, year 1 and year 2, all subsequent follow-up visits will be documented and entered into the JADE portal, which will then issue reports to both patients and doctor to promote sharing of information and informed decisions.
  Interventions: Other: JADE
- DIAMOND (Active Comparator): Patients will receive a comprehensive assessment at baseline, year 1 and year 2. In the interim between these time points patients will be managed according to 'usual care' procedures.
  Interventions: Other: DIAMOND

INTERVENTIONS:
Other: JADE — Patients are booked for reviews led by the doctor-nurse-HCA team every 2-4 months, preferably in a setting different from the busy clinics in order to facilitate group education and promote peer support.
  Between each follow-up visit, the nurse or HCA will contact the patient by phone or email to remind them of the appointments (e.g. medical FU visit or laboratory tests), adhere to medications and healthy lifestyles, perform self glucose monitoring and provide psychosocial support, as appropriate.
  Arms: JADE
Other: DIAMOND — Patients randomized to the DIAMOND group will receive usual care after the initial baseline comprehensive assessment (CA), with repeat CA at 12 and 24 months.
  Arms: DIAMOND

SUMMARY:
In this demonstration project (Asia Pacific JADE and DIAMOND Program, AP-JD in short) supported by the Asia Diabetes Foundation (ADF), patients will be recruited from different sites across Asia, with each site recruiting at least 600 type 2 diabetic patients. After explanation by trained doctors and nurses, and with written informed consent, patients will be randomized to either the JADE (n=300, structured care) or DIAMOND (n=300, usual care) group.

All patients will undergo a comprehensive assessment (CA) at baseline and yearly thereafter. Patients in the JADE group will be further managed by a doctor-nurse-HCA team according to a protocol based on risk stratification with predefined follow up (FU) schedules together with shared information and decision support (i.e. structured collaborative care). The DIAMOND protocol involves only baseline and yearly CA without predefined FU schedules or feedback of information between CA visits (i.e. usual care).

The primary composite endpoint is all-diabetes related clinical endpoints. The secondary composite endpoint is attainment of treatment goals and/or control of risk factors. The tertiary changes are behavioral changes, psychological well being and quality of life.

DETAILED DESCRIPTION:
Rationale: Change of practice environment and an interdisciplinary team is needed to implement evidence-based diabetes care which requires risk stratification, periodic assessments, education and treatment to targets.

Hypothesis: The use of a web-based disease management program (Joint Asia Diabetes Evaluation (JADE) Program) delivered by a doctor-nurse-HCA team reduces the incidence of all diabetes-associated clinical endpoint and improves control of risk factors compared to usual care (DIAbetes MONitoring Database (DIAMOND) group) in type 2 diabetes.

Objective: To compare structured care using the JADE portal versus usual care using the DIAMOND portal on incidence of all-diabetes related events, physical and psychological health.

Study design: A multicentre, randomized, integrated disease management program Setting and patients: 600 patients from each site will be randomized to the JADE group (n=300) or the DIAMOND group (n=300) and followed up for at least 24 months.

Intervention: All patients will undergo comprehensive assessment (CA) guided by the templates in the respective portal at baseline, month 12 and 24. The JADE group will be further managed by a doctor-nurse-HCA team guided by the JADE portal with risk stratification program and recommendation to different care protocols with predefined follow up (FU) schedules, information sharing and decision supports.

Outcome measures: Primary composite outcomes include all diabetes-related clinical events; secondary composite outcomes include control of risk factors and tertiary composite outcomes include behavioral changes, psychological health, quality of life and cost-effective analysis.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients who are willing or can be persuaded to return for 'regular' follow-up at 3-4 monthly intervals
* Patients with newly diagnosed or established disease, treated with lifestyle modification or blood glucose lowering drugs including oral agents with or without insulin
* For newly diagnosed type 2 diabetic patients, their plasma glucose levels should be:

  * Fasting plasma glucose (PG) >7.0 mmol/L on 2 or more occasions, and/or
  * Random or 2-hour PG >11.1 mmol/L (after 75 gram oral glucose tolerance test) on 2 or more occasions, and/or
  * HbA1c >6.5%

Exclusion Criteria:

* Type 1 diabetes defined as a history of ketosis at diagnosis [acute symptoms with heavy ketonuria (>3+) or ketoacidosis] or continuous requirement of insulin within one year of diagnosis
* Patients with reduced life expectancy (e.g. less than 6 months) due to recent diagnosis of advanced cancers (e.g. within last 2 years) and other life-threatening conditions
* Patients with a mental condition rendering them unable to understand the nature, scope, and possible consequences of the study
* Patients actively enrolled in another intervention study
* Patients who are unwilling to return for regular follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20834 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Incidence of all diabetes-related clinical endpoints | 12 months
  1. cardiovascular events (acute myocardial infarction, revascularisation procedures, heart failure, unstable angina, arrhythmia, stroke, transient ischemic attacks requiring hospital admissions)
  2. chronic kidney disease (eGFR<60 ml/min/1.73m2) or end stage renal disease (dialysis and/or eGFR<15 ml/min/1.73m2)
  3. visual impairment (corrected visual acuity of 20/200 or worse) or eye surgery
  4. lower extremity amputation or foot ulcers requiring hospitalizations
  5. major infections - pulmonary and non-pulmonary requiring hospitalizations
  6. all-site cancers
  7. death

SECONDARY OUTCOMES:
Proportions of patients with improved control of risk factors | 12 months
  a) 2 or more of the 'ABC' targets: i) HbA1c<7%, ii) BP<130/80 mmHg, iii) LDL-C <2.6 mmol/L.
  b) and/or
  c) 2 of the following changes in risk factor control: i) at least 0.5% reduction in HbA1c, ii) at least 5 mmHg reduction in systolic BP, iii) at least 0.5 mmol/L reduction in LDL-C, iv) at least 3% reduction in body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Chan, MD, Principal Investigator — Asia Diabetes Foundation
Locations (1):
- Asia Diabetes Foundation, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ko GT, So WY, Tong PC, Le Coguiec F, Kerr D, Lyubomirsky G, Tamesis B, Wolthers T, Nan J, Chan J. From design to implementation--the Joint Asia Diabetes Evaluation (JADE) program: a descriptive report of an electronic web-based diabetes management program. BMC Med Inform Decis Mak. 2010 May 13;10:26. doi: 10.1186/1472-6947-10-26. PMID 20465815
- [Background] Chan J, So W, Ko G, Tong P, Yang X, Ma R, Kong A, Wong R, Le Coguiec F, Tamesis B, Wolthers T, Lyubomirsky G, Chow P. The Joint Asia Diabetes Evaluation (JADE) Program: a web-based program to translate evidence to clinical practice in Type 2 diabetes. Diabet Med. 2009 Jul;26(7):693-9. doi: 10.1111/j.1464-5491.2009.02751.x. PMID 19573118
- [Derived] Lim LL, Lau ESH, Fu AWC, Ray S, Hung YJ, Tan ATB, Chamnan P, Sheu WHH, Chawla MS, Chia YC, Chuang LM, Nguyen DC, Sosale A, Saboo BD, Phadke U, Kesavadev J, Goh SY, Gera N, Huyen Vu TT, Ma RCW, Lau V, Luk AOY, Kong APS, Chan JCN; Asia-Pacific JADE Study Group. Effects of a Technology-Assisted Integrated Diabetes Care Program on Cardiometabolic Risk Factors Among Patients With Type 2 Diabetes in the Asia-Pacific Region: The JADE Program Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e217557. doi: 10.1001/jamanetworkopen.2021.7557. PMID 33929522
- See also: Asia Diabetes Foundation website — http://www.adf.org.hk